CLINICAL TRIAL: NCT06544980
Title: Measuring Upper Airway Cross Sectional Areas During Residual Neuromuscular Blockade and After Reserval
Status: Recruiting | Type: Observational
Sponsor: Tamas Vegh, MD (Other)
Responsible Party: Sponsor-Investigator, Tamas Vegh, MD, Head, Division of General, Vascular and Thoracic Anesthesia, University of Debrecen
Organization: University of Debrecen (Other)
Other Study IDs: AITT/2022/5; OGYEI/3962-11-/2023 (Other: National Institute of Pharmacy and Nutrition); DE RKEB/IKEB:625-2022 (Other: Regional and Institutional Ethics Committee University of Debrecen Clinical Center)
Record Dates: First submitted 2024-08-05; First posted 2024-08-09 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Postoperative Residual Curarization; Airway Obstruction on Anaesthetic Emergence
Keywords: residual neuromuscular blockade; postoperative airway obstruction; electromyography
MeSH Terms: conditions — Delayed Emergence from Anesthesia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In our study, the investigators sought to answer the question of how the retroglossal pharyngeal areas measured after extubation of patients compare to baseline (before muscle relaxation) values. The investigators also investigated how these areas change as a function of TOF ratios measured at extubation, thus looking for a correlation between residual muscle relaxant effect and airway area.

DETAILED DESCRIPTION:
Introduction

Postoperative residual neuromuscular can cause severe respiratory complications. One of these is pharyngeal dilator muscle weakness, which can lead to airway obstruction. One way to prevent this is to have objective neuromuscular monitors to track the degree of muscle relaxation and use the measurements to guide the the suspension of neuromuscular block. Monitoring the muscle relaxant effect is not a mandatory component of anaesthesia and is therefore often omitted in anaesthesiologists. In our study, the investigators investigated whether, at the end of surgery, only patients extubated at the end of surgery, based on clinical signs, have an airway diameter reduction and how this relates to the degree of residual muscle relaxation. Our single-centre, prospective study included 20 patients. The patients' narcosis by the anaesthetist, as is often done in routine anaesthesia work, is without monitoring neuromuscular block and on the basis of clinical signs deciding on extubation.

Sample size calculation

In a previous study, Eikermann and associates (Eikermann M, Vogt FM, Herbstreit F, Vahid-Dastgerdi M, Zenge MO, Ochterbeck C, de Greiff A, Peters J. The predisposition to inspiratory upper airway collapse during partial neuromuscular blockade. Am J Respir Crit Care Med. 2007;175(1):9-15.) using MRI technique described a minimal retroglossal diameter after a total neuromuscular recovery of 20.2±5.2 mm and a 20% decrease of this diameter at TOFR=0.8. the investigators hypothesised that in the present study, the decrease of the retroglossal cross-section area during inspiration will decrease by 30% in patients with residual neuromuscular block of any severity. Using and alpha of 0.05 and a power of 90%, 8 patients were calculated to be necessary to prove our hypothesis. In a previous study, it was found that in our working group the amount of residual neuromuscular block (as defined TOFR <90%) during spontaneous recovery at the end of surgery approximates 45% of all cases (Nemes R, Fülesdi B, Pongrácz A, Asztalos L, Szabó- Maák Z, Lengyel S, Tassonyi E. Impact of reversal strategies on the incidence of postoperative residual paralysis after rocuronium relaxation without neuromuscular monitoring: A partially randomised placebo controlled trial. Eur J Anaesthesiol. 2017;34(9):609-616.). With respect to this, the investigators planned to include 18 patients. the investigators also calculated with eventual dropouts and finally included 20 patients.

Procedure of the investigation

During the operation, the anaesthetist will routinely administer anaesthesia, including the selection of muscle relaxant and the timing of extubation. The latter is based solely on clinical signs and the anaesthetist performing narcosis does not use a neuromuscular monitor. However, the patients are not left without monitoring of the effect of the muscle relaxant, as an independent anaesthesiologist performs continuous electromyographic neuromuscular monitoring of the anaesthetised patients, the actual values of which are not known to the anaesthetist.

Medication of the patient, surgical procedure

As part of the balanced anaesthesia routinely used at the institute, the patient is first premedicated with 7.5 mg midazolam 60 minutes before the onset of anaesthesia. A peripheral vein is secured in one arm of the patient and infusion with Ringer's lactate solution is started. The other arm is left completely free for the independent anaesthetist, on which neuromuscular monitoring is performed throughout the operation. Continuous monitoring of the patient's physiological parameters is ensured by the use of precordial ECG, pulse oximetry, blood pressure measurement, central body temperature measurement, end-expiratory oxygen and CO2 measurement throughout the duration of the operation.

Induction of anaesthesia and maintenance of narcosis is achieved with total intravenous anaesthesia, propofol anaesthesia, TCI perfusion using the Schnider model. During induction, the propofol plasma concentration is set at 4-6 micrograms/ml. Before the administration of opioids and muscle relaxants, a control pharyngoscopy is performed, at which time the BIS index ranges between 60-70%. Patients are then asleep but spontaneous breathing is maintained. Once the recording is complete, the patient is given the type and dose of muscle relaxant chosen by the anaesthetist, fentanyl is administrated and the anethesist intubate the trachea. Subsequently, anaesthesia is deepened for the duration of the operation, with a BIS index of between 40-60%. The target concentration is then changed to 2.5-4 µg/ml to maintain narcosis. At the end of the operation, the non-monitoring anaesthetist performing the anaesthesia extubates the patient by observing the clinical signs, at which time the independent anaesthetist records the TOF value at the time of extubation. Fentanyl is antagonised while the patient is asleep. Pharyngoscopy is performed on the extubated patient. If necessary, i.e. when the TOF rate is below 90%, rescue medication is administered.

Neuromuscular monitoring

The anaesthetist did not monitor the patient, but the independent anaesthetist monitored the effects of the muscle relaxant throughout the operation. To do this, he uses a Tetragraph® electromyograph, which stimulates the ulnar nerve and detects the direct action potential of the adductor pollicis muscle. The application of the measuring instrument is facilitated by self-adhesive electrodes: the stimulating electrodes are placed on the volar surface of the wrist according to the course of the nerve mentioned above, and the sensing electrodes are placed towards the adductor pollicis muscle. The device is started with the patient already asleep, thus avoiding any discomfort due to stimulation. Once started, the device performs an autocalibration to determine the supramaximal excitation current to ensure muscle contraction. The electromyography uses the train of four -TOF stimulation pattern.

Offline analysis of pharnygoscopy and airway areas

During the examination of a patient, two pharyngoscopies are performed. The first one (called control pharnygoscopy) is performed under propofol but before the administration of opioid and muscle relaxant to ensure that the patient is breathing spontaneously. This is also to exclude the negative effect of opiate analgesia on the pharyngeal muscles. The second admission is performed after extubation. During the pharnygoscopy, a continuous chin lift, Escmarch-Heiberg manoeuvre, is used to guide the Ambu® aScope™ 4 Rhino Laryngo Slim rhino-laryngoscope down the nose to the vocal cord. The vocal fold was used as a landmark. From here, the camera was carefully retracted to locate the narrowest part of the pharynx, which corresponded to the retroglossal region. The found position is marked on the instrument with a marker, making it easier to find the same part of the pharynx for the second recording. During the pharyngoscopic examinations, moving images were also taken during the inhalation and exhalation phases, and these are analysed offline. Using the online available software Image J (Rasband WS, U.S. National Institutes of Health, Bethesda, Maryland, USA, https://imagej.net/ij/), the size of the airway areas is determined in pixels. From the resulting data set, the investigators can compare the data from control and end-of-operation pharyngoscopies and subsequently perform statistical calculations. Whenever possible, the investigators use analysis of variance (ANOVA) to estimate the parametric tests. Otherwise, the non-parametric Kruskal-Wallis test is used to compare each group. The significance level is defined as usual, p<0.05. Continuous variables are characterized by means and standard deviations.

Rescue medication

After pharyngoscopy, rescue medication is given if necessary, i.e. below 90% TOF, depending on the type of muscle relaxant used. If an aminosteroid muscle relaxant is used, the patient is given 2 mg/kg sugammadex, while if a benzylisoquinoline muscle relaxant is used, 0.05 mg/kg neostigmine and 0.015 mg/kg atropine are administrated to antagonise the drug effect.

ELIGIBILITY:
Inclusion Criteria:

Age: 18-65 years;

* ASA 1-3;
* BMI 18.5-25 (normal body weight);
* men/women in equal proportion;
* duration of surgeries at least ≥ 30 minutes;
* intervention requiring intratracheal intubation;
* patients are in a supine position.

Exclusion Criteria:

diseases affecting neuromuscular function (myopathies, severe liver and kidney failure);

* drugs affecting neuromuscular function (magnesium, aminoglycosides);
* difficult airway, expected difficult intubation;
* pregnancy (pregnancy test for women of childbearing age to rule out pregnancy we finish);
* breastfeeding;
* acute surgery;
* COPD
* glaucoma

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who receive a muscle relaxant (rocuronium bromide) for their operation to aid intubation and surgical exploration.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The differences in retroglossal pharyngeal cross sectional areas (inspiration and exspiration) measured at different TOF values | before intubation, after extubation of the trachea
  The differences in retroglossal pharyngeal cross sectional areas (inspiration and exspiration) measured at different train of four TOF values, and changes in these values compared to (initial) retroglossae pharyngeal areas detected before administration of muscle relaxants. Areas are measured in pixels and the rate of reduction of areas is expressed as a percentage.

CONTACTS AND LOCATIONS:
Overall Officials: László Asztalos, MD, PhD, Principal Investigator — Department of Anesthesiology and Intensive Care University of Debrecen
Locations (1):
- University of Debrecen, Debrecen, Hajdú-Bihar, Hungary

REFERENCES:
- [Background] Murphy GS, Szokol JW, Marymont JH, Greenberg SB, Avram MJ, Vender JS. Residual neuromuscular blockade and critical respiratory events in the postanesthesia care unit. Anesth Analg. 2008 Jul;107(1):130-7. doi: 10.1213/ane.0b013e31816d1268. PMID 18635478
- [Background] Ledowski T, Hillyard S, O'Dea B, Archer R, Vilas-Boas F, Kyle B. Introduction of sugammadex as standard reversal agent: Impact on the incidence of residual neuromuscular blockade and postoperative patient outcome. Indian J Anaesth. 2013 Jan;57(1):46-51. doi: 10.4103/0019-5049.108562. PMID 23716766
- [Background] Sundman E, Witt H, Olsson R, Ekberg O, Kuylenstierna R, Eriksson LI. The incidence and mechanisms of pharyngeal and upper esophageal dysfunction in partially paralyzed humans: pharyngeal videoradiography and simultaneous manometry after atracurium. Anesthesiology. 2000 Apr;92(4):977-84. doi: 10.1097/00000542-200004000-00014. PMID 10754616
- [Background] Arbous MS, Meursing AE, van Kleef JW, de Lange JJ, Spoormans HH, Touw P, Werner FM, Grobbee DE. Impact of anesthesia management characteristics on severe morbidity and mortality. Anesthesiology. 2005 Feb;102(2):257-68; quiz 491-2. doi: 10.1097/00000542-200502000-00005. PMID 15681938
- [Background] Eikermann M, Vogt FM, Herbstreit F, Vahid-Dastgerdi M, Zenge MO, Ochterbeck C, de Greiff A, Peters J. The predisposition to inspiratory upper airway collapse during partial neuromuscular blockade. Am J Respir Crit Care Med. 2007 Jan 1;175(1):9-15. doi: 10.1164/rccm.200512-1862OC. Epub 2006 Oct 5. PMID 17023729
- [Background] Herbstreit F, Peters J, Eikermann M. Impaired upper airway integrity by residual neuromuscular blockade: increased airway collapsibility and blunted genioglossus muscle activity in response to negative pharyngeal pressure. Anesthesiology. 2009 Jun;110(6):1253-60. doi: 10.1097/ALN.0b013e31819faa71. PMID 19417617
- [Background] Kirmeier E, Eriksson LI, Lewald H, Jonsson Fagerlund M, Hoeft A, Hollmann M, Meistelman C, Hunter JM, Ulm K, Blobner M; POPULAR Contributors. Post-anaesthesia pulmonary complications after use of muscle relaxants (POPULAR): a multicentre, prospective observational study. Lancet Respir Med. 2019 Feb;7(2):129-140. doi: 10.1016/S2213-2600(18)30294-7. Epub 2018 Sep 14. PMID 30224322
- [Background] Blobner M, Hunter JM, Meistelman C, Hoeft A, Hollmann MW, Kirmeier E, Lewald H, Ulm K. Use of a train-of-four ratio of 0.95 versus 0.9 for tracheal extubation: an exploratory analysis of POPULAR data. Br J Anaesth. 2020 Jan;124(1):63-72. doi: 10.1016/j.bja.2019.08.023. Epub 2019 Oct 10. PMID 31607388
- [Background] Heier T, Caldwell JE, Feiner JR, Liu L, Ward T, Wright PM. Relationship between normalized adductor pollicis train-of-four ratio and manifestations of residual neuromuscular block: a study using acceleromyography during near steady-state concentrations of mivacurium. Anesthesiology. 2010 Oct;113(4):825-32. doi: 10.1097/ALN.Ob013e3181ebddca. PMID 20808216
- [Background] Nemes R, Fulesdi B, Pongracz A, Asztalos L, Szabo-Maak Z, Lengyel S, Tassonyi E. Impact of reversal strategies on the incidence of postoperative residual paralysis after rocuronium relaxation without neuromuscular monitoring: A partially randomised placebo controlled trial. Eur J Anaesthesiol. 2017 Sep;34(9):609-616. doi: 10.1097/EJA.0000000000000585. PMID 28030444
- [Background] Fuchs-Buder T, Claudius C, Skovgaard LT, Eriksson LI, Mirakhur RK, Viby-Mogensen J; 8th International Neuromuscular Meeting. Good clinical research practice in pharmacodynamic studies of neuromuscular blocking agents II: the Stockholm revision. Acta Anaesthesiol Scand. 2007 Aug;51(7):789-808. doi: 10.1111/j.1399-6576.2007.01352.x. PMID 17635389
- [Background] Naguib M, Brull SJ, Kopman AF, Hunter JM, Fulesdi B, Arkes HR, Elstein A, Todd MM, Johnson KB. Consensus Statement on Perioperative Use of Neuromuscular Monitoring. Anesth Analg. 2018 Jul;127(1):71-80. doi: 10.1213/ANE.0000000000002670. PMID 29200077